CLINICAL TRIAL: NCT02410031
Title: Study to Evaluate Physician Knowledge of Safety and Safe Use Information for Diane-35 and Its Generics in Europe: An Observational Post-Authorisation Safety Study
Brief Title: Risk Minimisation Study for Diane-35 and Its Generics
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: RTI Health Solutions (Other)
Responsible Party: Sponsor
Other Study IDs: 17195
Record Dates: First submitted 2015-04-02; First posted 2015-04-07 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Cyproterone Acetate; Ethinyl Estradiol; Cyproterone acetate, ethinyl estradiol drug combination

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cyproterone acetate 2mg/ethinylestradiol 35 μg (Diane-35): Prescribers of Diane-35 who agree and fulfill the criteria inclusion to participate in the survey
  Interventions: Drug: Cyproterone acetate 2mg/ethinylestradiol 35 μg (Diane-35)

INTERVENTIONS:
Drug: Cyproterone acetate 2mg/ethinylestradiol 35 μg (Diane-35) — Cyproterone acetate 2mg/ethinylestradiol 35 μg

SUMMARY:
The study will be an observational, cross-sectional study of knowledge, understanding, and self-reported behavior among a sample of physicians with recent experience in prescribing Diane-35 or its generics in a total of five European countries. The primary objective of this study is to measure physician knowledge and understanding of the key information contained in the Diane-35 educational material: Patient information card, and Prescribers' Checklist.

Specifically, the following objectives will be addressed:

* Investigate whether physicians have received any educational material related to Diane-35 or its generics
* Assess physicians' knowledge and understanding of key safety information pertaining to the patient information card
* Assess physicians' knowledge and understanding of key safety information pertaining to the following areas:
* Contraindications relevant to thromboembolism
* Risk factors for thromboembolism
* Signs and symptoms of thromboembolism

ELIGIBILITY:
Inclusion Criteria:

-Physicians eligible to participate will have recently prescribed (e.g., within previous 6 months) Diane-35 or its generics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Physicians eligible to participate who have recently prescribed (e.g., within previous 6 months) Diane-35 or its generics
Sampling Method: Non-Probability Sample
Enrollment: 759 (Actual)
Dates: Start 2015-06-26 (Actual); Primary Completion 2016-03-04 (Actual); Study Completion 2016-03-04 (Actual)

PRIMARY OUTCOMES:
The knowledge of the physician concerning Diane-35 | Day1
  The knowledge will be assessed based on a questionnaire with 22 questions which wil assess physician knowledge on key information contained in the Diane-35 educational material including patient information card, prescribers' checklist

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (5):
- Many Locations, Austria
- Many Locations, Czechia
- Many Locations, France
- Many Locations, Netherlands
- Many Locations, Spain